CLINICAL TRIAL: NCT06353594
Title: Reduced Stent Strategy Versus Conventional Percutaneous Coronary Revascularization in Patients Presenting With St-segment Elevation Myocardial Infarction (Copernican)
Brief Title: Reduced Stent Strategy Versus Conventional Percutaneous Coronary Revascularization in Patients Presenting With STEMI
Acronym: COPERNICAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jorge Sanz Sanchez (Other)
Responsible Party: Sponsor-Investigator, Jorge Sanz Sanchez, Interventional cardiologist, Hospital Universitario La Fe
Organization: Hospital Universitario La Fe (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COPERNICAN TRIAL
Record Dates: First submitted 2024-03-14; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DCB-based (Experimental): Reduced stent PCI strategy: Culprit lesion revascularization with DCB will be performed after coronary predilation if residual stenosis ≤30%, lack of dissections >type B and TIMI 3 flow. If the aforementioned culprit-lesion characteristics are not achieved after DCB-PCI, a DES will be implanted.
  Interventions: Device: Primary PCI
- DES-based (No Intervention): Control group

INTERVENTIONS:
Device: Primary PCI — Coronary percutaneous revascularization
  Arms: DCB-based

SUMMARY:
The objective is to compare a reduced stent strategy based on drug-coated balloon (DCB) percutaneous coronary intervention (PCI) with conventional drug-eluting stent (DES) coronary revascularization in patients presenting with ST-segment myocardial infarction (STEMI).

Randomization will be performed after successful culprit-lesion guidewire crossing and flow restoration. Random allocation in a 1:1 fashion to one of the following strategies:

* Study group: reduced stent PCI strategy (DCB-based)
* Control group: conventional PCI strategy (DES-based).

ELIGIBILITY:
Inclusion Criteria:

- Patients presenting with STEMI and indication to undergo pPCI.

Exclusion Criteria:

* Life expectancy <1 year due 1 to non-cardiac disease.
* Inability to provide informed consent.
* Cardiogenic shock.
* Left ventricular ejection fraction <15%.
* Left main disease.
* Stent thrombosis
* Patients with prior bypass graft lesions requiring PCI (culprit or non culprit lesions).
* Patients with chronic total occlusions.
* Untreatable coronary disease.
* Non-identified culprit lesion.
* Known allergy to aspirin, ticagrelor, prasugrel, clopidogrel, paclitaxel or sirolimus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1272 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2035-09 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure (TLF) | 12 months
  Target-vessel myocardial infarction or ischemia-driven target-lesion revascularization

SECONDARY OUTCOMES:
Incidence of all-cause death | 10 years
  Physicians Assessment
Incidence of myocardial infarction | 10 years
  Physicians Assessment
Incidence of cardiovascular death | 10 years
  Physicians Assessment
Incidence of target lesion revascularization | 10 years
  Physicians Assessment
Incidence of stent thrombosis | 10 years
  Physicians Assessment
Incidence of acute vessel closure | 10 years
  Physicians Assessment
Incidence of stroke | 10 years
  Physicians Assessment
Incidence of acute kidney injury | 10 years
  Physicians Assessment
Incidence of bleeding | 10 years
  Physicians Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Sanz Sánchez, PI, Principal Investigator — Hospital Universitario La Fe; Ignacio J Amat Santos, PI, Principal Investigator — Hospital Universitario de Valladolid
Locations (15):
- Spain (15):
  - Hospital Universitario Y Politecnico La Fe, Valencia, Valencia
  - Consorcio Hospitalario Provincial de Castellon, Castelló
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Hospital Universitario Regional de Malaga, Málaga
  - Hospital Universitario de Navarra, Pamplona
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitari Joan Xxiii de Tarragona, Tarragona
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Hospital Clinico Universitario de Valladolid, Valladolid
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanz-Sanchez J, Santos Martinez S, Rumiz Gonzalez E, Oteo Dominguez JF, Tejada Ponce D, Gomez Menchero A, Sanchez Elvira G, Fuertes Ferre G, Rivero Crespo F, Lukic Otanovic A, Diaz Fernandez J, Galindo Fernandez E, Urbano Carrillo C, Salvatella Giralt N, Torres Sanchez M, Garcia Touchard A, Ibanez Cabeza B, Stefanini G, Alfonso Manterola F, Garcia Garcia H, Amat-Santos IJ. Reduced stent strategy versus conventional percutaneous coronary revascularization in patients presenting with STEMI: design of the COPERNICAN trial. Rev Esp Cardiol (Engl Ed). 2026 Feb;79(2):100-105. doi: 10.1016/j.rec.2025.05.005. Epub 2025 May 22. English, Spanish. PMID 40412715